CLINICAL TRIAL: NCT05357404
Title: Age and Sex-Specific PREValence of AcqUirEd VALVular Heart DiseasE (PREVUE-VALVE)
Brief Title: Age and Sex-Specific PREValence of AcqUirEd VALVular Heart DiseasE
Acronym: PREVUE-VALVE
Status: Active, not recruiting | Type: Observational
Sponsor: Cardiovascular Research Foundation, New York (Other)
Collaborators: CVS Caremark (Industry); Hawthorne Effect Inc. (Other); Columbia University (Other); Vanderbilt University Medical Center (Other); University of Michigan (Other); Walgreens (Industry)
Responsible Party: Sponsor
Other Study IDs: PREVUE VALVE
Record Dates: First submitted 2022-04-24; First posted 2022-05-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Valvular Heart Disease
Keywords: Valvular Heart Disease; Aortic Stenosis; Aortic Regurgitation; Mitral Regurgitation; Tricuspid Regurgitation; Epidemiology; Deep Learning; Electrocardiogram; Artificial intelligence; Biomarkers
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Study participants will have the option to undergo in-home phlebotomy in order to create a biospecimen repository ("biobank"). Blood samples will be collected during the home visit, and overnight mailed to the biobank core lab. Once they arrive at the biobank core lab, samples will be immediately processed, aliquoted, and frozen for future analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PREVUE-VALVE study will establish reliable, population-based estimates of Valvular Heart Disease (VHD) prevalence among older Americans and allow for the development and validation of several innovative tools to aid in the detection and diagnosis of Valvular Heart Disease (VHD).

DETAILED DESCRIPTION:
With the aging population, the incidence and prevalence of VHD are increasing in the U.S. and other parts of the developed world. Despite the availability of effective therapies and procedures to treat VHD, many patients remain (1) untreated due to undiagnosed VHD, or inadequate access to appropriate VHD care or (2) treated later than recommended due to diagnosis late in the disease course or barriers to prompt care for VHD. To optimize care for patients with VHD, it is therefore essential to (1) know the true prevalence of these conditions in order to align screening efforts with access to treatment; and (2) develop validated tools to more effectively screen and diagnose patients with VHD.

In response to these unmet needs, the PREVUE-VALVE study will establish reliable, population-based estimates of VHD prevalence in the United States and allow for the development and validation of several innovative tools to aid in the detection and diagnosis of VHD. The results of this study will enable the investigators to make tangible progress toward the goal of treating all patients with VHD at the optimal time.

The study will be conducted in a sample of older individuals (i.e., age 65-85 years) that is representative of the U.S. population. The sample will be carefully curated to ensure traditionally underrepresented individuals are included and overrepresented, if possible. After obtaining informed consent, each participant will undergo a standard echocardiogram in order to identify VHD (specifically aortic, mitral, and tricuspid valve disease) and to quantify its severity using state-of-the-art methods in a core echocardiography laboratory. Echocardiograms will be performed in participants' homes in an effort to reduce any barriers towards participation. A variety of complementary data (i.e. blood sample, electrocardiograms, and clinical inventory including a standardized health status assessment) will be collected while study personnel are with participants. Formal statistical weighting methods will be applied to estimate the population prevalence of various subtypes of VHD (e.g., aortic stenosis, mitral regurgitation) from the raw data. In addition, the investigators will report the prevalence of VHD, including VHD subtypes, and describe the association between different blood analytes and ECG characteristics with VHD.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-85
* Ability to provide informed consent
* Stably domiciled in a residence that can be accessed by study personnel

Exclusion Criteria:

* History of complex congenital heart disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults aged 65-85 will be eligible to participate. Population sampling techniques will be used to ensure that the study population is broadly representative of the age, sex, and racial distribution of the United States.
Sampling Method: Probability Sample
Enrollment: 2870 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Valvular Heart Disease | Baseline
  The primary endpoint of the study is the presence of any significant (i.e. moderate or greater) valvular heart disease at the baseline assessment including aortic stenosis, aortic regurgitation, mitral stenosis, mitral regurgitation, or tricuspid regurgitation.

SECONDARY OUTCOMES:
Moderate or greater aortic stenosis (at baseline) | Baseline
Moderate or greater aortic regurgitation (at baseline) | Baseline
Moderate or greater mitral stenosis (at baseline) | Baseline
Moderate or greater mitral regurgitation (at baseline) | Baseline
Moderate or greater tricuspid regurgitation (at baseline) | Baseline

OTHER OUTCOMES:
Descriptive Statistics | Baseline
  In addition to determining the population prevalence of each type of VHD at baseline, separate analyses will be performed to examine the cross-sectional relationship between age, sex, race, and ethnicity and the prevalence of valvular disease and its individual subtypes. The study will also evaluate the diagnostic performance of a machine learning model trained using 12-lead electrocardiograms to detect the primary endpoint and its components. Finally, the correlation between various blood analytes and significant valvular heart disease will also be assessed (specific analyses to be determined). In the future, long-term follow-up may be performed via linkage with health care claims data for patients who consent to this process.

CONTACTS AND LOCATIONS:
Overall Officials: David J Cohen, MD, Principal Investigator — CardioVascular Research Foundation
Locations (1):
- Hawthorne Effect, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No